CLINICAL TRIAL: NCT07317453
Title: Clinical Study for Precise Image for Musculoskeletal CT for Incisive CT and CT 5300 Systems
Brief Title: Precise Image for Musculoskeletal CT
Status: Not yet recruiting | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Collaborators: Philips Healthcare (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Precise Image for MSK
Record Dates: First submitted 2025-09-23; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-09

CONDITIONS: Computed Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
The purpose of this clinical study is to evaluate the performance of the Precise Image reconstruction algorithm for musculoskeletal CT imaging (shoulder, hip, knee) of adult patients (>18 years old). Clinical data generated from this study is intended to support a proposed expansion of the Indications for Use of Precise Image.

The study has two objectives:

1. To evaluate the image quality and diagnostic confidence of Precise Image compared to the standard-of-care reference (iDose4) for:

   * Musculoskeletal CT images (shoulder, hip, knee) of adult patients (>18 years old).
2. To demonstrate non-inferiority of Precise Image to iDose4 for the relevant resolution groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scanned by FDA-cleared and marketed Philips Incisive CT or CT 5300 systems, and according to the department standard of care clinical protocols for the applicable anatomies.
* Subject age: Above 18 years old.

Exclusion Criteria:

* Subject age: 18 years old and below.
* Scans that were acquired using generic 'Body' scan type (as Precise Image does not support generic 'Body' scan types).
* Scans that were acquired using a kilovoltage peak of 70 kVp (as Precise Image does not support a kilovoltage peak lower than 80 kVp).
* Scans that the site radiologists have deemed as non-diagnostic image quality in standard practice (e.g. patient movement).
* Scans that are not completed due to technical difficulties.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of CT Image quality and diagnostic confidence of Precise Image via 5-point Likert Scale | Reading session at 4 months
  The image quality and diagnostic confidence of Precise Image reconstructions is non-inferior to iDose4 reconstructions for musculoskeletal CT images of adult patients. Measurement will be done via 5-point Likert Scale for Image Quality where 5 is excellent and 1 is poor image quality.